CLINICAL TRIAL: NCT06795347
Title: Wellbeing and Resilience Among 1-3 Years Old Children of Mothers with Complex Mental Health Problems: a Pragmatic Clinical Trial
Brief Title: Wellbeing and Resilience Among 1-3 Years Old Children of Mothers with Complex Mental Health Problems: a Pragmatic Clinical Trial of Online VIPP-SD Vs. Care As Usual
Acronym: WellCom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kirstine Agnete Davidsen, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-20240007; 158789 (Other Grant/Funding Number: TrygFonden)
Record Dates: First submitted 2025-01-20; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Child Mental Health; Behavioral Symptoms; Child of Impaired Parents
Keywords: Parental psychiatric disorder; Child mental disorders; Prevention; Socio-emotional development; Child behavioral problems; Child externalizing problems; Parental sensitivity
MeSH Terms: conditions — Behavioral Symptoms; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (VIPP-SD) (Experimental): Video-feedback Intervention to promote Positive Parenting and Sensitive Discipline (VIPP-SD) delivered online
  Interventions: Behavioral: Online VIPP-SD
- Care As Usual (Other): Care As Usual is defined as any kind of help and support the parents may receive related to the socio-emotional development and mental wellbeing of their child in the municipality or the mental health services.
  Interventions: Behavioral: Care As Usual

INTERVENTIONS:
Behavioral: Online VIPP-SD — The Video-feedback Intervention to promote Positive Parenting and Sensitive Discipline is delivered online in this study. VIPP-SD is a manualized parenting intervention. The online version consists of 12 individual sessions, where the first and hereafter every second session consists of video recordings of mother and child in pre-defined everyday situations. The recordings are reviewed and discussed with the mother/parents during subsequent video-feedback sessions, where positive sequences in the interaction are pointed out by the intervener and form the basis of a discussion of pre-defined themes regarding child signals, attachment, child development, limit setting and sensitive parenting. The 12 sessions are conducted within five months from randomization with weekly or bi-weekly intervals.
  Arms: Intervention (VIPP-SD)
Behavioral: Care As Usual — Care As Usual is defined as any kind of help and support the parents may receive related to the socio-emotional development and mental wellbeing of their child in the municipality or the mental health services.
  Arms: Care As Usual

SUMMARY:
Children of parents with severe mental disorders have an increased risk of mental disorders themselves, with more than half of this population diagnosed with a mental health condition during their life time. Already during early childhood, the risk of a mental health diagnosis is elevated by a factor 2-5, compared to children of parents without severe mental disorders. This highlights the need for preventive interventions.

Mental health during early childhood is inextricably linked with early parent-child interaction. Sensitive parenting plays a crucial role in the socio-emotional development of the child, and severe parental mental disorders may affect the quality of parent-child interaction.

Therefore, we will test the effect of an intervention promoting sensitive parenting on mental health outcomes of 1-3 years old children of parents with severe mental disorders. The intervention will be tested in a randomized clinical trial comparing the intervention "Video-feedback Intervention to Promote Positive Parenting and Sensitive Discipline" (VIPP-SD) delivered online to Care As Usual. Our hypothesis is, that children in the Intervention Group will display lower levels of behavioral problems and increased attachment security compared to children in the Care As Usual Group.

The study will be conducted in the department of Child and Adolescent Psychiatry, Mental Health Services in the Region of Southern Denmark. Participants are mothers with a diagnosis of schizophrenia, bipolar disorder, emotionally unstable personality disorder or moderate to severe depression living in the Region of Southern Denmark with their 1-3 years old child, and the father/cohabitating partner. Participants will be recruited via psychiatric outpatient clinics in the region or on the basis of information from health registers.

The primary outcome of the study is child behavioral problems. Secondary child outcomes are attachment security and mental health. Parental outcomes are parental stress and quality of life. Child cognition, parental psychiatric symptoms, childhood trauma, sensitivity, parental reflective functioning and service use data are also assessed in the study. Data are collected at baseline as well as 5 and 11 months after randomization. All participants will have the opportunity to receive feedback on their child's cognitive functioning and mental health status at baseline and at the end of the study.

After baseline assessments, participants will be randomized to either intervention or the control group.

The intervention, VIPP-SD, is delivered online apart from the first session, which is conducted as a home visit. VIPP-SD is based on attachment and social learning theory. It is manualized and consists of 12 individual sessions alternating between video-recording of mother and child in pre-defined everyday situations and review/discussion of the video recordings with the mother/parents. Focus of the intervention is the childs signals and needs, and how to promote healthy socio-emotional development of the child. VIPP-SD will be carried out by health care professionals trained and certified in VIPP-SD.

Participants who are randomized to the control condition, Care As Usual, will continue as they did before enrollment to the study. Care As Usual is defined as any kind of help and support related to the social-emotional development and mental wellbeing of the child in the municipality or mental health services.

ELIGIBILITY:
Inclusion Criteria:

* child age 1 year, 0 months until 3 years, 0 months
* living with their mother in the Region of Southern Denmark
* mother has a mental disorder (Schizophrenia ICD-10: F20-29, Bipolar disorder ICD-10: F30-31, Moderate to severe depression ICD-10: F32-33 or Emotionally unstable personality disorder F60.3) verified in the Danish National Hospital Register-Psyk/the Danish Psychiatric Central Research Register or by a clinician at the mental health services via the patient record
* mother has had at least one in- or outpatient contact with mental health services within 12 months before birth of the child or during the child's lifetime verified in the Danish National Hospital Register or by a clinician at the mental health services via the patient record

Exclusion Criteria:

* current in-patient status of the mother
* current substance or alcohol abuse of the mother
* mother has insufficient knowledge of Danish (interpreter required)
* repeated intrauterine exposure to euphoriants or large amounts of alcohol (≥5 units per time or ≥7units per week) of the child
* known syndrome or autism spectrum disorder of the child
* mother or child has sensory impairment
* sibling participating in study
* family participating in another closely related research trial receiving an individualized video-feedback intervention
* participating in active court proceedings

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Preschool Parental Account of Children's symptoms (P-PACS) | The P-PACS will be administered at baseline (T0), 5 months (T1) and 11 months (T2) after randomization.
  The P-PACS is a semistructured researcher-led interview administered to the mother, assessing level of child behavioral problems. Change in level of child behavioral problems is the primary outcome of the study.

SECONDARY OUTCOMES:
Child Behavior Check List/1 ½-5 (CBCL/1 ½-5) | CBCL/1 ½-5 will be administered at baseline (T0), 5 months (T1) and 11 months (T2) after randomization.
  The Danish version of the CBCL/1 ½-5 will be completed by both (cohabitating) parents. Change in Total problems score, and Internalizing and Externalizing subscale scores is used as a secondary outcome measure.
Caregiver-Teacher Report Form (C-TRF) | C-TRF will be administered at baseline (T0), 5 months (T1) and 11 months (T2) after randomization.
  The Danish version of the C-TRF will be completed by the child's day care teacher. Change in Total problems score, and Internalizing and Externalizing subscale scores is used as a secondary outcome measure.
Baby-DIPS | Baby-DIPS will be administered at baseline (T0), 5 months (T1) and 11 months (T2) after randomization.
  The Baby-DIPS is a structured interview designed for the diagnosis of former and current regulatory problems (excessive crying, feeding or sleeping disorder). It is conducted with the mother. Change in regulatory problems will be used as a secondary outcome.
the Brief Attachment Scale-16 (BAS-16) | The BAS-16 will be administered at baseline (T0) and 11 months (T2) after randomization.
  BAS-16 is used for evaluating child attachment security in relation to both mother and (cohabitating) father. The BAS-16 is based on two scales, the "happy and harmonious interactions" and "proximity and physical-contact seeking". Change in mean score will be used as outcome.
Parental Stress Scale (PSS) | The Parental Stress Scale will be administered at baseline (T0), 5 months (T1) and 11 months (T2) after randomization.
  The questionnaire Parental Stress Scale will be completed by both (cohabitating) parents. A total score and two subscale scores (Parental Stress and Parental Satisfaction) will be calculated.
  Change in mean scores will be used as outcome.
Parental Sensitivity | Sensitivity will be assessed at T0 and T1.
  Parental sensitivity wil be assessed with the Coding of Interactive behavior on the basis of video-recordings of child in interaction with mother and father/cohabitating partner during a structured interaction containing a difficult task. The sensitivity socre is a composite score based on predefined parental subscales and ranges between one and five, with high scores indicating a high degree of sensitivity.
Parental Reflective Functioning Questionnaire (PRFQ) | The PRFQ will be completed by both (cohabitating) parents at baseline (T0), 5 months (T1) and 11 months (T2) after randomization.
  The PRFQ is a questionnaire assessing self-reported parental reflective functioning. The items are divided into three categories: Prementalizing modes, Certainty about mental states and Interest and curiousity about mental states.
EQ-5D-5L | EQ-5D-5L will be administered at baseline (T0), 5 months (T1) and 11 months (T2) after randomization.
  Quality of life is assessed with the Danish version of the EQ-5D-5L, a self-report measure assessing the impact of health on an individual's everyday life. EQ-5D-5L is completed by both (cohabitating) parents. Change in mean score will be used as secondary outcome measure.
Symptom Checklist-90-revised (SCL-90-R) | The SCL-90-R is completed at baseline (T0), 5 months (T1) and 11 months (T2) after randomization.
  The SCL-90-R is a self-report questionnaire, which will be used to evaluate parental psychopathology. It is completed by both (cohabitating) parents.

CONTACTS AND LOCATIONS:
Overall Officials: Davi, Principal Investigator — Region of Southern Denmark
Locations (1):
- Research Unit of Child and Adolescent Psychiatry, Mental Health Services in the Region of Southern Denmark, Odense C, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No